CLINICAL TRIAL: NCT05014243
Title: Targeted Metabolomics to Decipher Dietary Contributions to Pediatric Inflammatory Bowel Disease (IBD)
Brief Title: Targeted Metabolomics to Decipher Dietary Contributions to Pediatric Inflammatory Bowel Disease (IBD) - Main Study
Acronym: TAMED IBD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 20-0369
Record Dates: First submitted 2021-05-21; First posted 2021-08-20 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Gut Microbiome; Inflammation; Irritable Bowel Syndrome
MeSH Terms: conditions — Inflammation; Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Stool and urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The overall goal of the study is to investigate the dietary differences between children with well-controlled inflammatory bowel disease (IBD) and those with active disease by using targeted food metabolomics. The utilization of the application of targeted metabolomics allows for the investigation of specific components of foods and their effects in IBD and inflammation, which may inform future dietary recommendations for IBD patients.

DETAILED DESCRIPTION:
The investigators overall hypothesis is that higher intake of animal origin foods lead to higher concentrations of TMAO and its precursors (TMA, choline and carnitine), which causes gut microbiota dysbiosis, ultimately resulting in elevated inflammatory markers (systemic and/or fecal) in pediatric inflammatory bowel disease (IBD).

The two primary aims include:

Aim 1: Examine the relationship between IBD activity, dietary patterns, and diet-derived potential biomarkers in serum and urine.

Aim 2: Investigate the association between IBD activity, dietary patterns, gut microbiome, and diet-derived potential biomarkers in stool.

Investigators will also explore the integrated relationship between disease activity, diet, gut microbiome, diet-derived potential biomarkers, and inflammatory markers.

Investigators will recruit 100 subjects with known IBD of > 6 months duration. Subjects will be asked to complete dietary questionnaires, and provide stool, urine, and blood samples.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female
* Established IBD diagnosis (both well-controlled and active disease) for > 6 months
* Followed by the Children's Hospital Colorado (CHCO) IBD Center
* Ages 8-18 years

Exclusion Criteria:

* Vegan diet
* Exclusive enteral nutrition (EEN) currently or within 2 weeks of enrollment
* History of full colectomy
* Ongoing active gastrointestinal infection
* Severe malnutrition (BMI less than 5th percentile)
* Presence of ostomy
* Recent medication changes

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with established IBD diagnosis (both well-controlled and active disease) for > 6 months
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Diet-derived potential biomarkers | Collected within 4 weeks of consent
  Serum, urine, and stool concentrations of TMAO, TMA, choline and carnitine
Dietary Intake - 24 Hour Food Recall | Collected within 4 weeks of consent
  The Automated Self-Administered 24-Hour (ASA24®) Dietary Assessment is used to collect recall and food record data and measures healthy eating and overall diet quality. Macronutrient composition and mean intake will be reported.
Dietary Intake - BLOCK Questionnaire for Ages 8-17 - 2004 FFQ | Collected within 4 weeks of consent
  BLOCK includes 77 food items. Individual portion size is asked, and pictures are provided to enhance accuracy of quantification. BLOCK will be analyzed for each subject and raw data for nutrient intake. The number of servings of food groups will be assessed, and specific nutrient intake will be calculated and reported as mean intake.
Fecal microbiome | Collected within 4 weeks of consent
  Deep shotgun sequencing to assess the gut microbiome
Inflammatory markers | Collected within 4 weeks of consent
  Erythrocyte sedimentation rate (ESR), C-reactive protein (CRP) and calprotectin

IPD SHARING:
Plan to Share IPD: No